CLINICAL TRIAL: NCT02445300
Title: Efficacy of Wound Care and Reduction of Wound Complications by Use of AQUACEL® Ag Surgical Dressing in Minimally Invasive Total Knee Arthroplasty：A Prospective, Randomized Controlled Study
Brief Title: Efficacy of Wound Care and Reduction of Wound Complications by Use of AQUACEL® Ag Surgical Dressing in MIS TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Feng Chih Kuo, Feng Chih Kuo, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMPRG8C0711
Record Dates: First submitted 2015-04-14; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Complication
Keywords: dressing; TKA
MeSH Terms: conditions — Postoperative Complications | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AQUACEL® Ag Surgical dressing (Active Comparator): AQUACEL® Ag Surgical dressing is used to cover the surgical wound in the OR. Clinical indications for removal of the AQUACEL® Ag Surgical dressing were leakage from the dressing beyond the hydrocolloid exterior layer and more than a 50% saturation of the Hydrofiber® inner layer.
  Interventions: Other: AQUACEL® Ag Surgical dressing (study group)
- Sofra-Tulla® dressing (Active Comparator): The Sofra-Tulle® dressing was used in the OR and routinely changed at a daily basis. If there were strikethrough on the gauze, the nursing staff would proceed the dressing change automatically between the daily routine.
  Interventions: Other: Sofra-Tulle® dressing (control group)

INTERVENTIONS:
Other: AQUACEL® Ag Surgical dressing (study group) — The AQUACEL® Ag Surgical dressing was applied to the wound in the operating theater by the surgeon. Clinical indications for removal of the AQUACEL® Ag Surgical dressing were leakage from the dressing beyond the hydrocolloid exterior layer and more than a 50% saturation of the Hydrofiber® inner layer10. If there were no indications to change the dressing, it was changed at the day of discharge usually the 4th or 5th postoperative day (POD) and remained cover of the wound for 7 days except for exudate across the dressing.
  Arms: AQUACEL® Ag Surgical dressing
Other: Sofra-Tulle® dressing (control group) — The Sofra-Tulle® dressing was applied to the wound in the operating theater by the surgeon. The Sofra-Tulle® dressing was routinely changed at a daily basis. If there were strikethrough on the gauze, the nursing staff would proceed the dressing change automatically between the daily routine. After discharge from the hospital, the family who had been taught well to do this job during the patient's stay in the hospital conducted the daily dressing change.
  Arms: Sofra-Tulla® dressing

SUMMARY:
The investigators hypothesized that AQUACEL® Ag Surgical dressing would have a significant improvement in the efficacy of wound care and wound complications compared with traditional Sofra-Tulle® dressings after minimally invasive total knee arthroplasty (MIS-TKA).

DETAILED DESCRIPTION:
Traditional adhesive dressing (Mepore®; Mölnlycke Health Care) for low limb arthroplasty wounds had blistering up to 26%. The jubilee dressing, which consisted of a highly absorbent Hydrofiber inner layer and (Aquacel; ConvaTec Inc.) and a viscoelastic hydrocolloid outer layer (DuoDERM Extra Thin; ConvaTec Inc.), was introduced for lower limb arthroplasty wounds with lower blistering rate (2% vs. 18%) and lower surgical site infection (1% vs. 3%) compared to traditional adhesive dressing. A new modern dressing regime (Aquacel Ag Surgical dressing; ConvaTec Inc.) also reported longer wear time, less dressing change and less blistering.

In our institution, the standard wound care after TKA was an antimicrobial dressing (Sofra-Tulle®; Royal Chem. & Pharm. Co., Kaohsiung, Taiwan) in the inner layer and gauzes in the outer layer.

The investigators hypothesized that AQUACEL® Ag Surgical dressing would have a significant improvement in the efficacy of wound care and wound complications compared with traditional Sofra-Tulle® dressings after MIS-TKA.

ELIGIBILITY:
Inclusion Criteria:

* Two hundred and eighty five patients who were scheduled for primary unilateral MIS-TKA were enrolled in the study period.

Exclusion Criteria:

* Patients with condition/comorbidity that could compromise wound healing, including varicose eczema, peripheral vascular disease, receiving immunosuppressive medications, corticosteroid abuse, chronic skin disease around the knee (e.g. psoriasis and chronic eczema) and having prior knee replacement, osteotomy or fracture of the ipsilateral knee.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Wound Care Efficacy | an expected average of 5 days at the duration of hospital stay
  Wear time, No. of dressing change,
Number of Participants with Adverse Events | Three months after surgery
  Blister formation, wound erythema, discharge and necrosis
ASEPSIS score | 2 weeks after surgery
  Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissue, Isolation of bacteria and Stay as inpatient
Surgical site infection (SSI) | Three months after surgery
  Superficial or deep infection of the wound

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | two weeks after surgery
  overall pain management, and removal when using the dressings
Comfort scale | two weeks after surgery
  The dressing is comfort in use and ease of application (excellent, good, fair or poor)
Ease scale | two weeks after surgery
  The dressing is ease of application and removal (excellent, good, fair or poor)

CONTACTS AND LOCATIONS:
Overall Officials: FENG-CHIH KUO, MD, Study Chair — Chang Gung Memorial Hospital